CLINICAL TRIAL: NCT05686486
Title: Impact of a Joint Practice of a Tai Chi Inspired Gymnastics Program on the Relationship Between Family Caregivers and Residents in Nursing Homes
Brief Title: Gentle Gymnastics and Relationship Between Family Caregivers and Residents With Dementia in Nursing Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondation Mederic Alzheimer (Other)
Collaborators: Malakoff-Humanis (Unknown); Siel Bleu (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FMAR-010; ID RCB : 2021-A02651-40 (Other: French ANSM)
Record Dates: First submitted 2023-01-03; First posted 2023-01-17 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2023-03

CONDITIONS: Dementia; Relation, Family
Keywords: Dementia; Nursing homes; Psychosocial intervention; Family relationship; Family caregivers
MeSH Terms: conditions — Dementia

STUDY DESIGN:
Intervention Model Description: The experimental design is a cluster randomised controlled study with three arms corresponding to three experimental conditions. Sixty dyads will be recruited for a total of 120 participants (60 family caregivers and 60 residents) divided into 12 groups.
  9 nursing homes are participating.
Who Masked: Outcomes Assessor
Masking Description: Investigators, participants and professionals are aware of the experimental condition. Only the external evaluators do not know which experimental condition the participants are in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Tai Chi inspired gymnastics practiced in a family caregiver-resident dyad (residents) (Experimental): 15 participants in 3 groups with 5 residents per group who benefited with 5 family caregivers from the Tai Chi inspired gymnastics programme at a rate of two one-hour sessions per week for 12 weeks.
  Interventions: Other: Tai Chi inspired gymnastics
- Tai Chi inspired gymnastics practised individually (residents) (Active Comparator): 30 participants in 3 groups with 10 residents per groups who benefited separately from the family caregivers from the Tai Chi inspired gymnastics programme at a rate of two one-hour sessions per week for 12 weeks.
  Interventions: Other: Tai Chi inspired gymnastics
- Control group (residents) (No Intervention): 15 participants in 3 groups with 5 residents. As well as their family carers, they did not benefit from the intervention the study. They will be able to continue their usual activities. At the end of the study, they will be offered the 24 sessions of the Tai Chi inspired gymnastics programme in family caregiver-resident dyad.
- Tai Chi inspired gymnastics practiced in a family caregiver-resident dyad (family caregivers) (Experimental): 15 participants in 3 groups with 5 family caregivers per group who benefited with 5 residents from the Tai Chi inspired gymnastics programme at a rate of two one-hour sessions per week for 12 weeks.
  Interventions: Other: Tai Chi inspired gymnastics
- Tai Chi inspired gymnastics practised individually (family caregivers) (Active Comparator): 30 participants in 3 groups with 10 family caregivers per groups who benefited separately from the residents from the Tai Chi inspired gymnastics programme at a rate of two one-hour sessions per week for 12 weeks.
  Interventions: Other: Tai Chi inspired gymnastics
- Control group (family caregivers) (No Intervention): 15 participants in 3 groups with 5 family caregivers. As well as the residents, they did not benefit from the intervention the study. They will be able to continue their usual activities. At the end of the study, they will be offered the 24 sessions of the Tai Chi inspired gymnastics programme in family caregiver-resident dyad.

INTERVENTIONS:
Other: Tai Chi inspired gymnastics — The intervention programme will address the themes of "relax and seek flexibility" and "contact and follow". The programme will be divided into four parts with six sessions per part. A typical session will be as follows:
  * Joint warm-up
  * A body session focused on relaxation and flexibility in different planes: sagittal/sagittal and frontal/sagittal, frontal and transversal/sagittal, frontal and transversal.
  * A more playful session in pairs on the theme of "contact and follow". Example: put the back of your hand against the back of your partner's hand and initiate movements and the other must follow without resistance.
  Arms: Tai Chi inspired gymnastics practiced in a family caregiver-resident dyad (family caregivers); Tai Chi inspired gymnastics practiced in a family caregiver-resident dyad (residents); Tai Chi inspired gymnastics practised individually (family caregivers); Tai Chi inspired gymnastics practised individually (residents)

SUMMARY:
The goal of this multicentre cluster randomised controlled trial is to evaluate the effects of a joint practice of a Tai Chi inspired gymnastics programme in nursing home on the relationship between family caregivers and residents living with mild to moderate dementia. The intervention consists of 24 sessions of Tai Chi inspired gymnastics programme for two one-hour sessions per week in a family caregiver-resident pair. The researchers will compare the practice of the intervention in pairs with a separate practice and with the absence of intervention to see if any effects are observed on the family caregiver-resident relationship. The hypotheses are as follows:

* Hypothesis 1: the relationship between family caregiver and resident will be judged better after the joint practice of a Tai Chi inspired gymnastics programme compared to a separate practice and compared to no intervention.
* Hypothesis 2: signs of anxiety and depression in the family caregiver and resident should be lower after joint practice of a Tai Chi inspired gymnastics programme compared to separate practice and compared to no intervention.
* Hypothesis 3: the family caregivers' feeling of competence will be higher after the joint practice of a Tai Chi inspired gymnastics programme compared to a separate practice and compared to no intervention.
* Hypothesis 4: the quality of life of the residents will be better after the joint practice of a Tai Chi inspired gymnastics programme compared to a separate practice and compared to no intervention.

DETAILED DESCRIPTION:
An information letter was sent to nursing homes in the Lille region (France) to present the objectives of the study. The nursing homes that agreed to participate received additional information for implementing the study. Randomisation was carried out in clusters, i.e. the sites were randomised to one of the three experimental conditions. The randomisation was carried out using Excel (Microsoft Corporation, version 18.2110.13110.0). For each site, a random value was generated and then a rank was assigned for each value. The rank value was divided by three, corresponding to the number of experimental conditions. These values were then rounded up. Each site therefore has a value of "1", "2" or "3" corresponding to an experimental condition: "1" = arm #1; "2" = arm #2; and "3" = arm #3.

The investigators of the 9 participating nursing homes screened the residents and family caregivers according to inclusion, non-inclusion and exclusion criteria. The study was then presented to residents and family caregivers who met the criteria by giving them an information letter so that they could take time to consider whether to participate in the study, with a minimum two-week cooling-off period between the information and the written consent.

The socio-demographic data collected will concern for all participants: age; gender; level of education; relationship in the dyad; previous practice of Tai Chi; usual sports and leisure activities. For residents, the Mini Mental State Examination (MMSE) score will also be collected from the medical record of each included resident and must be less than six months old. If the MMSE score is older than six months, the nursing homes will be asked to carry out the MMSE.

Two assessments of the residents and family caregivers will be carried out before the intervention and two weeks after the intervention. The assessments will be carried out by psychologists who have been previously informed and/or trained in the use of the questionnaires and scales. The information and/or training will be done by telephone. Evaluations will be conducted blind, i.e. psychologists will not be aware of the experimental condition that will be assigned to each participant. Each evaluation will last between 30 minutes and 1 hour.

Data collection in the observation books will be carried out via a code assigned to each participant in a non-identifying manner. A table of correspondence between the participants' first and last names and the codes will be kept securely by the principal investigator at each site. Once the data collection is finalised, these tables will be deleted and the codes will not appear on the computer files used for data processing and statistical analysis.

Data will be stored in each nursing home for the duration of the study. Only authorised principal investigators will have access to the consent forms and observation books for the duration of the study, which will be anonymised. The external evaluators will have access to the observation books via by the principal investigators of each sites only during the evaluations.

The coordinating investigator will make monitoring visits to ensure the proper implementation of the study and the accuracy of the consent and data collection. The coordinating investigator will also be in regular contact by email and telephone with the principal investigator at each site.

The results of the tests and scales will be processed descriptively and analysed statistically with comparisons of means between the three experimental conditions. The results will also be analysed taking into account signs of anxiety, depression and the quality of the caregiver-caregiver relationship before the start of the study. The qualitative data will be analysed for content.

ELIGIBILITY:
Inclusion Criteria for the residents:

* Agreement of the resident and the family caregiver to participate in the study;
* Presence of neurocognitive disorders mentioned in the resident's file and objectified by a MMSE score between 16 and 25 out of 30;
* Presence in the nursing home for more than six months;
* Ability to attend the sessions;
* Ability to walk to the place of the intervention alone, with human or technical assistance.
* Medical advice indicating the possibility of practising the activity.

Exclusion Criteria for the residents:

* Refusal of the resident or of the family caregiver to continue the study;
* Alteration of the general state of health no longer allowing participation in the sessions and assessments;
* Hospitalization(s) that do not allow regular follow-up of the sessions and evaluations;
* Permanent leaving of the nursing home;
* Death.

Inclusion Criteria for the family caregivers:

* Medical certificate by the general practitioner indicating the possibility of carrying out the Tai Chi inspired gymnastics sessions;
* Family caregiver having frequent contact with the resident: spouse; child; brother/sister; cousin;
* Agreement of the family caregiver and the resident to participate in the study;
* Absence of neurocognitive disorders;
* Ability to attend the proposed sessions;
* Operational mobility to go to the intervention site.

Exclusion Criteria for the family caregivers:

* Refusal of the family caregiver or of the resident to continue the study;
* Alteration of the general state of health no longer allowing participation in the sessions and assessments;
* Hospitalization(s) that do not allow regular follow-up of the sessions and evaluations;
* Death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2023-02-06 (Actual); Study Completion 2023-02-06 (Actual)

PRIMARY OUTCOMES:
Questionnaire of relationship between family caregivers and residents - Residents' point of view | Baseline
  A 12-questions questionnaire will assess the family caregiver-resident relationship from the perspective of the residents. For each question, the residents will choose from four answers the one that is closest to what they think at the time of the questionnaire, e.g. "You think about your relative: all the time, often, rarely, never". Each question is rated from 0 to 3 for a maximum score of 36. A high score indicates a good perceived relationship. The questions are the same for family caregivers and residents to calculate a final relationship score by averaging the family caregiver's score and the resident's score. Additional questions not included in the score of relationship are asked to assess the relationship qualitatively.
Questionnaire of relationship between family caregivers and residents - Residents' point of view questionnaire | 2 weeks after the intervention
  A 12-questions questionnaire will assess the family caregiver-resident relationship from the perspective of the residents. For each question, the residents will choose from four answers the one that is closest to what they think at the time of the questionnaire, e.g. "You think about your relative: all the time, often, rarely, never". Each question is rated from 0 to 3 for a maximum score of 36. A high score indicates a good perceived relationship. The questions are the same for family caregivers and residents to calculate a final relationship score by averaging the family caregiver's score and the resident's score. Additional questions not included in the score of relationship are asked to assess the relationship qualitatively.
Questionnaire of relationship between family caregivers and residents - Family caregivers' point of view | Baseline
  A 12-questions questionnaire will assess the family caregiver-resident relationship from the perspective of the family caregivers. For each question, the family caregivers will choose from four answers the one that is closest to what they think at the time of the questionnaire, e.g. "You think about your relative: all the time, often, rarely, never". Each question is rated from 0 to 3 for a maximum score of 36. A high score indicates a good perceived relationship. The questions are the same for family caregivers and residents to calculate a final relationship score by averaging the family caregiver's score and the resident's score. Additional questions not included in the score of relationship are asked to assess the relationship qualitatively.
Questionnaire of relationship between family caregivers and residents - Family caregivers' point of view | 2 weeks after the intervention
  A 12-questions questionnaire will assess the family caregiver-resident relationship from the perspective of the family caregivers. For each question, the family caregivers will choose from four answers the one that is closest to what they think at the time of the questionnaire, e.g. "You think about your relative: all the time, often, rarely, never". Each question is rated from 0 to 3 for a maximum score of 36. A high score indicates a good perceived relationship. The questions are the same for family caregivers and residents to calculate a final relationship score by averaging the family caregiver's score and the resident's score. Additional questions not included in the score of relationship are asked to assess the relationship qualitatively.

SECONDARY OUTCOMES:
Hospital Anxiety and Depression Scale (HAD) | Baseline and 2 weeks after the intervention
  This scale consists of 14 items and two subscales of seven items each: a subscale assessing anxiety and a subscale assessing depression.This scale is administered to residents and family caregivers.The maximum score on each subscale is 21. A score of 7 or less indicates no symptomatology; a score between 8 and 10 indicates probable symptomatology; and a score of 11 or more indicates certain presence of symptomatology.
Sense of Competence Questionnaire (QSC) | Baseline and 2 weeks after the intervention
  This questionnaire consists of 27 items describing how one feels about helping a person living with dementia through three aspects: satisfaction with one's own performance as a caregiver, the consequences for the caregiver's personal life and the satisfaction given to the caregiver by the patient.This questionnaire is administered to family caregivers.The maximum score is 27. The higher the score, the better the feeling of competence.
Quality of Life-Alzheimer's Disease scale in Nursing Homes (QOL-AD NH) | Baseline and 2 weeks after the intervention
  This scale assesses the perceived quality of life of residents living in nursing home with mild to moderate Alzheimer's disease or a related disorder (MMSE ≥10/30). This scale can be analysed globally and across three dimensions: quality of life related to the intra- and interpersonal environment; quality of life related to personal functioning; and quality of life related to current perceived health.This scale is administered to the residents.The total score is between 15 and 60. The higher the score, the higher the perceived quality of life.
Mini Mental State Examination (MMSE) | Baseline
  This test was designed for the rapid detection and monitoring of cognitive deficits. The MMSE will be administered to family caregivers prior to the start of the intervention to ensure that there is no cognitive impairment.This test is scored out of 30 points and consists of 6 categories: temporo-spatial orientation (10 points), 3-word learning (3 points), attention-calculation (5 points), 3-word recall (3 points), language (8 points) and constructive praxis (1 point).

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Bernard Mabire, PhD, Principal Investigator — Fondation Mederic Alzheimer
Locations (4):
- France (4):
  - Résidence Les Terrasses de la Scarpe, Courchelettes
  - EHPAD Afeji Edilys, Lille
  - EHPAD Korian Samara, Marpent
  - EHPAD Afeji Les Tilleuls, Maubeuge

IPD SHARING:
Plan to Share IPD: No